CLINICAL TRIAL: NCT05211180
Title: Vida Sana y Completa Trial: Treating Obesity and Food Insecurity Among Latina Women
Brief Title: Vida Sana y Completa Obesity and Food Insecurity Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); San Mateo Medical Center (Other)
Responsible Party: Principal Investigator, Lisa Goldman Rosas, Principal Investigator, Assistant Professor, Department of Health Research and Policy (Epidemiology) and Medicine (Primary Care and Population Health) Faculty Director, Office of Community Engagement Stanford School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 63206
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: obesity; food insecurity; Latina; fitbit; Metabolic Diseases; Chronic Disease
MeSH Terms: conditions — Obesity; Metabolic Diseases; Chronic Disease

STUDY DESIGN:
Intervention Model Description: This study uses a type 1 hybrid design with participants randomized in a 1:1 ratio to either Vida Sana y Completa (an obesity intervention with integrated treatment for food insecurity) or Vida Sana alone (the comparator arm). Vida Sana is a cultural-adaption of Group Lifestyle Balance, a 12-month intervention that targets at least 5% weight loss and at least 150 minutes per week of moderate-to-vigorous physical activity.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will know which group they have been randomized to. The investigator and statistician will not know which group a participant belongs to. Group identifiers will be removed prior to analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vida Sana (Active Comparator): Vida Sana is a cultural-adaption of Group Lifestyle Balance, a 12-month intervention that targets at least 5% weight loss and at least150 minutes per week of moderate-to-vigorous physical activity. Health coaches will facilitate 12 weekly 1-hour group education sessions, followed by nine 30-45 minute individual monthly phone sessions. Health coaches will also conduct two home visits (at baseline and 12-weeks post-enrollment). The health coach will review participant's fitbit health tracking data with them and give personalized feedback.
  Interventions: Behavioral: Vida Sana
- Vida Sana y Completa (Experimental): Vida Sana y Completa is an obesity intervention with integrated treatment for food insecurity. This arm includes all the activities described for the active comparator arm (Vida Sana) as well as a weekly food box delivery for the first 12 weeks of the intervention. The food box will contain approximately 40 pounds of food including proteins and dairy, whole grains, and produce. Just like the Vida Sana active comparator arm, the Vida Sana y Completa group will include health coaches who will facilitate 12 weekly 1-hour group education sessions, followed by nine 30-45 minute individual monthly phone sessions. Health coaches will also conduct two home visits (at baseline and 12-weeks post-enrollment). The health coach will review participant's fitbit health tracking data with them and give personalized feedback.
  Interventions: Behavioral: Vida Sana y Completa

INTERVENTIONS:
Behavioral: Vida Sana — Weekly group or individual education sessions with a health coach and fitness tracking with a fitbit.
  Arms: Vida Sana
Behavioral: Vida Sana y Completa — Weekly group or individual education sessions with a health coach, fitness tracking with a fitbit, and weekly food box delivery.
  Arms: Vida Sana y Completa

SUMMARY:
The goal of the Vida Sana y Completa study is to provide evidence on the most effective approach for addressing the critical combination of obesity and food insecurity among Latinas in primary care while also collecting preliminary information on the potential for implementation and dissemination.

DETAILED DESCRIPTION:
The goal of this study is to compare two approaches to addressing obesity and food insecurity among Latina women in primary care to provide evidence for community health centers who serve this high-priority group. The project team will recruit 412 low-income Latina women with obesity (body mass index 30) and food insecurity from two community health centers with whom the team has longstanding partnerships. Patients will be randomized to Vida Sana y Completa (an obesity intervention with integrated treatment for food insecurity) or Vida Sana alone. Vida Sana is a state-of-the-art cultural adaptation of Group Lifestyle Balance, a 12-month program that targets at least 5 percent weight loss and at least 150 minutes per week of moderate-to-vigorous physical activity. For food insecurity, the team will provide boxes of healthy foods (e.g., fresh produce, lean protein, low-fat dairy, and whole grains) that give women the foods they need to adopt a healthy diet.

ELIGIBILITY:
Inclusion Criteria:

* Age: Lower age limit - 18 years, Upper age limit - NONE
* Race/ethnicity: self-reported Latinx ethnicity
* Sex: Female
* Body mass index: ≥ 30 kg/m2
* One or more metabolic risk factors as follows:
* Fasting plasma glucose of 100 to 125 mg/dL or HbA1c of 5.7 to 6.4 if detected by a recent (within the past year), documented, blood-based diagnostic test in the Electronic Health Record (EHR) in the last year
* Waist circumference >40 inches in men and >35 inches in women (≥35 inches in men and ≥31 inches in women, if of Asian descent) as measured by the study coordinator
* Triglycerides >150 mg/dL as documented in the EHR in the last year
* High-density lipoprotein cholesterol (HDL-C) <40 mg/dL in men and <50 mg/dL in women as documented in the EHR in the last year
* Systolic blood pressure >120 mmHg or diastolic blood pressure >80 mmHg as measured by study coordinator
* Food insecurity: Defined as answering yes to one or both questions of the Hunger Vital Sign
* PCP approval of patient contact for study screening
* Able and willing to enroll and provide informed consent, i.e., to meet the time and data collection requirements of the study, be randomized to one of 2 study arms, participate for 24 months, and authorize extraction of relevant information from the EHR.

Exclusion Criteria:

* Previous diagnosis of diabetes (other than during pregnancy) or diabetes documented in the EHR
* Diagnosis of cancer (other than non-melanoma skin cancer) that is/was active or treated with radiation or chemotherapy within the past 2 years
* Serious medical condition anticipated to prevent person from walking

  1 mile (e.g., severe pulmonary disease or aortic stenosis)
* Severe medical comorbidities that require aggressive treatment: e.g., stage 4 or greater renal disease, class III or greater heart failure, unstable coronary artery disease, liver or renal failure;
* Diagnosis of a terminal illness and/or in hospice care;
* Diagnosis of bipolar disorder or psychotic disorder within the last 2 years, or currently taking a mood stabilizer or antipsychotic medication
* Initiation or change in type or dosing of antidepressant medications within 2 months prior to enrollment (The patient will be re-contacted for a later cohort once his/her regimen has been stable for at least 2 months unless the person declines to participate altogether.)
* Have had or plan to undergo bariatric surgery during the study period

Other exclusions:

* Inability to speak, read or understand Spanish
* Having no reliable telephone service
* Having no regular Internet access via a computer and/or mobile device (e.g., smartphone)
* Plan to move out of the area during the study period
* Planned pregnancy
* Family/household member of another study participant or of a study staff member
* Investigator discretion for clinical safety or protocol adherence reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Weight change (12 months) | Baseline, 12 months, 24 months
  Trained research assistants blinded to treatment assignment will weigh participants in duplicate using a standard calibrated scale at baseline, 12, and 24 months

SECONDARY OUTCOMES:
Self-reported weight | 6 months, 18 months
  Participants will self-report measures of weight at 6 and 18 months to the health coach via telephone.
Visit or EHR Height, Weight, and Waist Circumference | baseline, 12 months, 24 months
  In person visits at baseline, 12-months and 24-months post enrollment will be used to collect participant weight, height and waist circumference. At baseline, these will be measured twice or in triplicate if there is a discrepancy. Height will be measured in centimeters, weight will be measured in kilograms, and waist circumference will be recorded in centimeters. If participants cannot be weighed in person for the primary outcome, weight measurement from the EHR if available within 3 months of the data collection date will be used.
  Waist circumference will be measured according to standard protocols described by the National Health and Nutrition Examination Surveys (NHANES) Anthropometry Procedures Manual. http://www.cdc.gov/nchs/data/nhanes/nhanes_11_12/Anthropometry_Procedures_Manual.pdf. Published 2011.
Health-related quality of life | baseline, 6 months, 12 months, 24 months
  The validated SF-8™ will be used. It is a generic multipurpose short-form health-related quality of life instrument and was developed by the RAND Corporation and the Medical Outcomes Study (MOS) in the 1980s.
Obesity-specific quality of life | baseline, 6 months, 12 months, 24 months
  Obesity-related Problem Scale, average scores of 8 questions with a range from 0 (no at all) to 3 (extremely). The average score is then multiplied by 100 and divided by 3 to convert to a scale of 0-100, with a higher score indicating more obesity-related problems. Obesity-related quality of life measured at baseline, 6 months, 12 months and at 24 months.
Change in Psychosocial Well-being: Depressive Symptoms | baseline, 6 months, 12 months, 24 months
  The Patient Health Questionnaire PHQ-9 is a self-report questionnaire with 9 items plus a 10th question. Respondents answered questions regarding how often a symptom has bothered them over the last two weeks. Each item is rated on a 4-point scale (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day). PHQ-9 total score is the sum of the nine items, ranging from 0 to 27. Scores of 5, 10, 15, and 20 represent cut-points for mild, moderate, moderately severe and severe depression, respectively. PHQ-9 score at baseline, 6 months, 12 months and at 24 months.
Cardiometabolic risk factors | baseline, 6 months, 12 months, 24 months
  Waist circumference will be measured at baseline, 12 months and at 24 months according to standard protocols described by the National Health and Nutrition Examination Surveys (NHANES) Anthropometry Procedures Manual. http://www.cdc.gov/nchs/data/nhanes/nhanes_11_12/Anthropometry_Procedures_Manual.pdf. Published 2011. Accessed October 29, 2014.
  At baseline, 12 months and at 24 months blood pressure will be measured twice by a trained health coach, a third if there is a discrepancy. Blood pressure, fasting glucose, HbA1c, and lipids will be pulled from the medical record for each time point.
Participant Medication Usage | baseline, 12 months, 24 months
  Participants will be asked to self-report medications/prescriptions. A list of prescribed medications will also be pulled from the electronic health record.
Dietary Intake Patterns | baseline, 6 months, 12 months, 24 months
  Dietary intake will be measured using the gold-standard approach of 3 multiple pass 24-hour recalls (2 during the weekday and 1 on the weekend at each time point). The Nutrition Data System for Research (NDSR), a validated approach, will be used. Changes in dietary intake over 24-months will be assessed.
Food Neophobia Scale | baseline, 6 months, 12 months, 24 months
  The Food Neophobia Scale (FNS) is a 10-item questionnaire that is comprised of likert type items ranging from "strongly disagree (1)" to "strongly agree (7)." Participants indicate their level of agreement for statements such as "I will eat almost anything" with higher scores indicating greater agreement per item.
Food Attitudes & Behaviors (FAB) Scale for self-efficacy | baseline, 6 months, 12 months, 24 months
  A subset of 7 items regarding Self-Efficacy to Eat Fruits and Vegetables will be used from the validated Food Attitudes & Behaviors (FAB) scale. These items are answered on a likert scale from "not at all confident" to "very confident" with an option for "does not apply." Scoring details are available on the NIH website (https://cancercontrol.cancer.gov/brp/hbrb/food-attitudes-and-behaviors).
Second Harvest of Silicon Valley Food Bank Self-Efficacy Measure | baseline, 6 months, 12 months, 24 months
  Two self-reported items from the Second Harvest of Silicon Valley food bank self-efficacy questionnaire will be asked. They are "In the past few months, have you tried a new recipe using food you received at a free food distribution?" and "And have you tried a new fruit or vegetable that you received at a free food distribution?" Answer choices are yes, no, or I did not receive food.
Participant self-reported 7-day Physical Activity Recall | baseline, 6 months, 12 months, 24 months
  The research team will administer the 7-day Physical Activity Recall, a self-report measure of physical activity and sleep.
Participant steps per day | baseline, 6 months, 12 months, 18 months, 24 months
  Steps per day will be verified with data from the Fitbit Alta HR used to calculate steps per day.
Number of participants with food insecurity | baseline, 6 months, 12 months, 18 months, 24 months
  The USDA 6-item brief food security measure is a validated tool for assessing household food security. Food security status for each participant at 5 time points over 24 months will be recorded.
Self-reported Nutrition Security, Healthfulness Control, and Utilization Barriers Survey Tool | baseline, 6 months, 12 months, 18 months, 24 months
  Each participant self-report answers 4 self-report nutrition security questions, 2 questions about control over the food consumed, and 2 questions about barriers over the last 12 months. Answers choices are a likert scale from Never=0 to Always=4 with higher scores indicating lower levels of nutritional security.
  Sample item: "In the last 12 months, (I/we) had to eat some foods that were not good for (my/our) health and well-being because (I/we) could not get other types of food."
Stunkard Figure Rating Scale | baseline
  Motivation for weightloss will be measured using the Stunkard Figure Rating Scale. This validated tool uses a diagram showing figures of various shapes and sizes and asks the participant to indicate their current body type and the type they would most like to be. Participants are asked to: (1) choose your ideal figure; (2) choose the figure that reflects how you think you look; (3) choose the figure that reflects how you feel most of the time; (4) choose the figure that you think is most preferred by men; (5) choose the figure that you think is most preferred by women; and (6) pick the opposite sex figure that you find most attractive. Scoring uses discrepancy measures: (1) feel minus ideal; (2) think minus ideal; and (3) feel minus think
  Thompson, J.K., & Altabe, M.N. (1991). Psychometric qualities of the figure rating scale. International Journal of Eating Disorders, 10(5), 615-619.
Level of anxiety among participants | baseline, 6 months, 12 months, 24 months
  The validated Generalized Anxiety Scale (GAD-7) will be administered to measure the severity of anxiety that may be present among participants. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 indicate mild, moderate and severe anxiety, respectively.
Bidimensional Acculturation Scale for Hispanics | baseline
  This validated self-report 24-item tool will be used to understand how participants communicate in both English and Spanish. Each item is a likert-type with answer choices asking participants to rate the frequency they use a communication practice. Answers range from "Almost always (4)" to "Almost never (1)" or "Very well (4)" to "Very Poorly (1)."
COVID-19 Impact on Health and Wellbeing Survey for Health Literacy | baseline
  Four items were selected from the COVID-19 Impact on Health and Wellbeing Survey to capture how participants receive and process health information such as level of comfort with health forms, medical information, and visiting the doctor.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Goldman Rosas, PhD, MPH, Principal Investigator — Stanford University; Wei-ting Chen, PhD, Study Director — Stanford University
Locations (1):
- San Mateo Medical Center Fair Oaks Health Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers

REFERENCES:
- [Background] Straub SX, Garry RF, Magee WE. Interferon induction by poly (I): poly (C) enclosed in phospholipid particles. Infect Immun. 1974 Oct;10(4):783-92. doi: 10.1128/iai.10.4.783-792.1974. PMID 4426708
- [Background] Conzelmann E, Sandhoff K. The specificity of human N-acetyl-beta-D-hexosaminidases towards glycosphincolipids is determined by an activator protein. Adv Exp Med Biol. 1980;125:295-306. doi: 10.1007/978-1-4684-7844-0_27. PMID 6444774
- [Background] Copeland MM. American Joint Committee on Cancer Staging and end results reporting. Objectives and progress. Cancer. 1965 Dec;18(12):1637-40. doi: 10.1002/1097-0142(196512)18:123.0.co;2-c. No abstract available. PMID 5845801
- [Background] Pliner P, Hobden K. Development of a scale to measure the trait of food neophobia in humans. Appetite. 1992 Oct;19(2):105-20. doi: 10.1016/0195-6663(92)90014-w. PMID 1489209
- [Background] Thompson, J.K., & Altabe, M.N. (1991). Psychometric qualities of the figure rating scale. International Journal of Eating Disorders, 10(5), 615-619.
- See also: Food Attitudes and Behaviors (FAB) from NIH — https://cancercontrol.cancer.gov/brp/hbrb/food-attitudes-and-behaviors
- See also: National Health and Nutrition Examination Surveys (NHANES) Anthropometry Procedures Manual — http://www.cdc.gov/nchs/data/nhanes/nhanes_11_12/Anthropometry_Procedures_Manual.pdf.